CLINICAL TRIAL: NCT04992117
Title: Unplanned-extubation in the Intensive Care Unit; Incidence, Characteristics and Prognosis.
Brief Title: Unplanned-extubation in the ICU; Incidence, Characteristics and Prognosis. Success And Failure of Self-Extubation in the ICU
Acronym: SAFE-ICU
Status: Completed | Type: Observational
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: SAFE-ICU / NR-2021-02
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Unplanned Extubation; Self Extubation
Keywords: Self extubation; Unplanned extubation; intensive care unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unplanned-extubation in the ICU: Patients with unplanned extubation in the ICU
  Interventions: Other: NO INTERVENTION

INTERVENTIONS:
Other: NO INTERVENTION — NO INTERVENTION

SUMMARY:
Our study consists of a national observational study assessing quantitatively (incidence) and qualitatively unscheduled extubation in intensive care unit. In addition, we will compare the outcome of patients with "success" or "failure" in the self-extubation subgroup.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Mechanically ventilated with oral or nasotracheal intubation
* Occurrence of an unscheduled extubation (auto-extubation or accidental extubation)
* Extubation is defined as the removal of the orotracheal or nasotracheal tube with the impossibility of reinsertion of the same device.

Exclusion Criteria:

* Opposition to the use of personal data
* Pregnant women
* Person under protective custody or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with occurrence of an unscheduled extubation (auto-extubation or accidental extubation) in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 633 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Quantitative description | During stay in the ICU
  Quantitative description of unscheduled extubation episodes in intensive care unit

SECONDARY OUTCOMES:
Qualitative description | During stay in the ICU
  Qualitative description of unscheduled extubation episodes in intensive care unit
re-intubation | During stay in the ICU
  To assess factors associated with re-intubation
Severe hemodynamic and respiratory events | One hour after extubation
  To assess the incidence of severe hemodynamic and respiratory events of immediate onset
Length of stay in intensive care unit, the duration of mechanical ventilation and mortality | During stay in the ICU
  Compare the length of stay in intensive care unit, the duration of mechanical ventilation as well as the mortality in intensive care of subjects with "successful self-extubation" (defined as no re-intubation on D7) compared to those in "failure of" self-extubation ".

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel CONSTANTIN, MD, Study Chair — Hôpital La Pitié Salpêtrière - Paris
Locations (1):
- Hôpital La Pitié Salpêtrière- Département d'Anesthésie-Réanimation, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided